CLINICAL TRIAL: NCT05753501
Title: First-in-Human Study to Evaluate the Safety, Pharmacokinetics, and Preliminary Efficacy of the BTK Degrader, ABBV-101, in Participants With B-cell Malignancies
Brief Title: Study to Evaluate Adverse Events, Change in Disease Activity, and How Oral ABBV-101 Moves Through the Body in Adult Participants With B-Cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M23-647; 2023-503594-38-00 (Other: EU CT)
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hematologic Cancer
Keywords: Chronic lymphocytic leukemia (CLL); Small lymphocytic lymphoma (SLL); Chimeric antigen receptor T-cells (CAR-T); Hematopoietic cell transplant (HCT); Relapsed/refractory (R/R) or ineligible Diffuse large b-cell lymphoma (DLBCL); Mantle cell lymphoma (MCL); Follicular lymphoma (FL); Marginal zone lymphoma (MZL); Waldenström macroglobulinemia (WM); Transformed Indolent non-Hodgkin's lymphoma (INHL); Hematologic Cancer; ABBV-101
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Escalation ABBV-101 (Experimental): Participants with relapsed or refractory (R/R) Non-Hodgkin's lymphoma (NHL) will receive escalating doses of ABBV-101, until the maximum administered dose (MAD)/Maximum tolerated dose (MTD) is determined, as part of the approximately 88 month study duration.
  Interventions: Drug: ABBV-101
- Dose Expansion ABBV-101 R/R CLL/SLL (Experimental): Participants with R/R chronic lymphocytic lymphoma (CLL)/small lymphocytic lymphoma (SLL) will receive ABBV-101 at the dose determined in the dose escalation arm, as part of the approximately 88 month study duration.
  Interventions: Drug: ABBV-101
- Dose Expansion ABBV-101 R/R non-GCB DLBCL (Experimental): Participants with R/R non-germinal center B cell (GCB) diffuse large B-cell lymphoma (DLBCL) will receive ABBV-101 at the dose determined in the dose escalation arm, as part of the approximately 88 month study duration.
  Interventions: Drug: ABBV-101

INTERVENTIONS:
Drug: ABBV-101 — Oral:Tablet

SUMMARY:
Non-Hodgkin's lymphoma (NHL) is a cancer that arises from the transformation of normal B and T lymphocytes (white blood cells). The purpose of this study is to assess the safety, pharmacokinetics, and preliminary efficacy of ABBV-101 in adult participants in relapsed or refractory (R/R) non-Hodgkin's lymphomas: chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), diffuse large b-cell lymphoma (DLBCL), non-germinal center B cell (GCB) DLBCL, mantle cell lymphoma (MCL), follicular lymphoma (FL), marginal zone lymphoma (MZL), Waldenström macroglobulinemia (WM), or transformed indolent NHL. Adverse events will be assessed.

ABBV-101 is an investigational drug being developed for the treatment of NHL. This study will include a dose escalation phase to determine the maximum administered dose (MAD)/Maximum tolerated dose (MTD) of ABBV-101 and a dose expansion phase to determine the change in disease activity in participants with first line treatment (1L), second line or later of treatment (2L)+ CLL/SLL or third line or later of treatment (3L) non-GCB DLBCL. Approximately 340 adult participants with multiple NHL subtypes will be enrolled in the study in sites world wide.

In the Dose Escalation phase of the study participants will receive escalating oral doses of ABBV-101, until the MAD/MTD is determined, as part of the approximately 88 month study duration. In the dose expansion phase of the study participants receive oral ABBV-101, as part of the approximately 88 month study duration .

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, and side effects.

ELIGIBILITY:
Inclusion Criteria:

* For Dose Escalation (Part 1) only: Participants have received at least two prior systemic therapies, have no available therapies known to provide clinical benefit (e.g., standard chemotherapy or HCT), have measurable disease requiring treatment, and have a documented diagnosis for one of the following third line or later B-cell malignancies, from one of the following world health organization (WHO)-defined histologies (Swerdlow et al 2016):

  * Chronic lymphocytic leukemia (CLL)
  * Small lymphocytic lymphoma (SLL)
  * Chimeric antigen receptor T-cells (CAR-T)/hematopoietic cell transplant (HCT) relapsed/refractory (R/R) or ineligible diffuse large b-cell lymphoma (DLBCL) from the following histologies: DLBCL not otherwise specified (NOS) (germinal center B cell [GCB] and non-GCB DLBCL), T-cell/histiocyte-rich large B-cell lymphoma, primary mediastinal (thymic) large B-cell lymphoma, intravascular large B-cell lymphoma, anaplastic lymphoma kinase positive (ALK+) large B-cell lymphoma, high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements, and high-grade B-cell lymphoma NOS.
  * Mantle cell lymphoma (MCL)
  * Follicular lymphoma [FL] (grades 1-3b)
  * Marginal zone lymphoma [MZL] (splenic, extranodal, and nodal)
  * Waldenström macroglobulinemia (WM)
  * Transformed indolent non-Hodgkin's lymphoma (iNHL)

    1. For Dose Escalation (Part 1) - BTKi/BTKd-naïve CLL/SLL backfill only: Participants with a documented diagnosis of CLL/SLL who have received at least one prior systemic therapy that cannot be a BTK inhibitor or degrader, and, with the exception of BTK pathway agents, have no available therapies known to provide clinical benefit (e.g., standard chemotherapy or HCT), and have measurable disease requiring treatment.
    2. For Dose Escalation (Part 1) - BTKi/BTKd-naïve CLL/SLL backfill only: Participants with a documented diagnosis of CLL/SLL who have received one prior systemic therapy with a BTKi and BCL-2i combination regimen, have no available therapies known to provide clinical benefit (e.g., standard chemotherapy or HCT), and have measurable disease requiring treatment.
* For Dose Expansion (Part 2) CLL/SLL only: Participants with a documented diagnosis of CLL/SLL who have received at least one prior systemic therapy.
* For Dose Expansion (Part 2) DLBCL only: Participants have received at least two prior systemic therapies, have no available therapies known to provide clinical benefit (e.g., standard chemotherapy or HCT), have measurable disease requiring treatment, and have a documented diagnosis of CAR-T/HCT R/R or ineligible non-GCB DLBCL in their third line or later treatment with histology based on criteria established by the World Health Organization (WHO).
* Has an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0, 1, or 2. For EU only: Participant has an ECOG PS of 0 or 1.
* Participant has a life expectancy >= 12 weeks.
* Prior Bruton's tyrosine kinase inhibitor (BTKi) is allowed.
* Adequate hematologic, renal, and hepatic function per the protocol.

Exclusion Criteria:

* Previously treated with a Bruton's tyrosine kinase (BTK) degrader.
* Known active central nervous system (CNS) disease, or primary CNS lymphoma. Participants with prior CNS disease that have been effectively treated may be eligible.
* Uncontrolled active systemic infection requiring systemic treatment that is ongoing or was completed <= 14 days before the first dose of study drug, or active cytomegalovirus infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AE) | Up to Approximately 88 Months
  AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Change in Laboratory Parameters | Up to Approximately Two Years
  Number of participants with clinically significant change from baseline in clinical laboratory test results like hematology will be reported.
Change in Vital Signs | Up to Approximately Two Years
  Number of participants with clinically significant change from baseline in vital signs like systolic and diastolic blood pressure will be reported.
Change in Electrocardiogram (ECG) | Up to Approximately Two Years
  12-lead resting ECGs will be recorded. Parameters include RR interval, PR interval, QT interval, and QRS duration.

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of ABBV-101 | Up to Approximately One Year
  Maximum observed serum concentration of ABBV-101.
Time to Cmax (Tmax) of ABBV-101 | Up to Approximately One Year
  Time to Cmax of ABBV-101.
Area Under the Serum Concentration Versus Time Curve (AUC) of ABBV-101 | Up to Approximately One Year
  Area under the serum concentration versus time curve (AUC) of ABBV-101.
Number of Participants with Response of Partial Response (PR) or Better Response (Overall Response) per Disease-Specific Criteria | Up to Approximately Two Years
  Number of participants with response of PR or better response (overall response) per disease-specific criteria.
Duration of Response (DOR) | Up to Approximately Two Years
  DOR is defined for participants achieving PR or better as the time from the initial response per Investigator review to disease progression or death of any cause, whichever occurs earlier.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (51):
- United States (14):
  - Arizona Oncology Associates, PC-HOPE /ID# 252351, Tempe, Arizona
  - UC Irvine Medical Center /ID# 263020, Orange, California
  - Stanford University /ID# 249683, Palo Alto, California
  - Rocky Mountain Cancer Centers - Lone Tree /ID# 252237, Lone Tree, Colorado
  - Northwestern University Feinberg School of Medicine /ID# 249347, Chicago, Illinois
  - Beth Israel Deaconess Medical Center /ID# 249302, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey /ID# 249323, New Brunswick, New Jersey
  - New York Oncology Hematology - Albany Cancer Center /ID# 252240, Albany, New York
  - Northwell Health - Monter Cancer Center /ID# 250422, Lake Success, New York
  - University of Rochester Medical Center /ID# 249324, Rochester, New York
  - UC Health - Cincinnati /ID# 249299, Cincinnati, Ohio
  - Oncology Assoc. of Oregon PC - WVCI and Research Ctr - Springfield /ID# 249309, Eugene, Oregon
  - University of Pennsylvania /ID# 250341, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center /ID# 249293, Houston, Texas
- Canada (2):
  - University Health Network_Princess Margaret Cancer Centre /ID# 253483, Toronto, Ontario
  - CHUM Notre-Dame Hospital /ID# 253428, Montreal, Quebec
- France (6):
  - Institut Bergonie /ID# 253664, Bordeaux, Gironde
  - CHU Montpellier - Hopital Saint Eloi /ID# 253666, Montpellier, Herault
  - CHRU Lille - Hopital Claude Huriez /ID# 253665, Lille, Nord
  - Centre Hospitalier Universitaire de Nantes, Hotel Dieu -HME /ID# 256248, Nantes, Pays de la Loire Region
  - Institut Gustave Roussy /ID# 253662, Villejuif, Val-de-Marne
  - Hôpital Saint-Louis /ID# 253663, Paris
- Germany (6):
  - Universitaetsklinikum Ulm /ID# 253742, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Wuerzburg /ID# 254636, Würzburg, Bavaria
  - Universitaetsmedizin Rostock /ID# 259657, Rostock, Mecklenburg-Vorpommern
  - Universitaetsklinikum des Saarlandes /ID# 257435, Homburg, Saarland
  - Charite Universitaetsklinikum Berlin - Campus Benjamin Franklin /ID# 257431, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 264566, Hamburg
- Israel (4):
  - Yitzhak Shamir Medical Center /ID# 254566, Ẕerifin, Central District
  - Hadassah Medical Center-Hebrew University /ID# 251123, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 251122, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 259608, Tel Aviv, Tel Aviv
- Italy (5):
  - IRCCS Ospedale San Raffaele /ID# 253531, Milan, Milano
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 253532, Milan, Milano
  - A.O.U. CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO - Ospedale Molinette /ID# 253530, Turin, Piedmont
  - ASST Papa Giovanni XXIII /ID# 260317, Bergamo
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 255172, Bologna
- Japan (4):
  - National Cancer Center Hospital East /ID# 250684, Kashiwa-shi, Chiba
  - Kyoto University Hospital /ID# 261837, Kyoto, Kyoto
  - National Cancer Center Hospital /ID# 250680, Chuo-ku, Tokyo
  - The Cancer Institute Hospital Of JFCR /ID# 260375, Koto-ku, Tokyo
- Spain (6):
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 260196, Majadahonda, Madrid
  - Hospital Universitario Vall de Hebron /ID# 260447, Barcelona
  - Hospital Universitario Ramon y Cajal /ID# 260450, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 253654, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 253655, Madrid
  - Hospital Universitario de Salamanca /ID# 253656, Salamanca
- United Kingdom (4):
  - Addenbrookes Hospital /ID# 256242, Cambridge, Cambridgeshire
  - Leicester Royal Infirmary /ID# 255171, Leicester, England
  - University College London Hospital /ID# 260202, London, Greater London
  - Kings College Hospital NHS Foundation Trust /ID# 253670, London, Greater London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related info — https://www.abbvieclinicaltrials.com/study/?id=M23-647